CLINICAL TRIAL: NCT06445686
Title: Ongoing Monitoring of Vital Signs in Patients With Idiopathic Pulmonary Fibrosis Before and After Acute Exacerbation. (REACT)
Brief Title: Ongoing Monitoring of Vital Signs in Patients With Idiopathic Pulmonary Fibrosis Before and After Acute Exacerbation.
Acronym: REACT
Status: Recruiting | Type: Observational
Sponsor: Biosency (Industry)
Collaborators: Rennes University Hospital (Other); Air de Bretagne (Unknown); Association Fibroses Pulmonaires France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2023-A02063-42
Record Dates: First submitted 2024-05-29; First posted 2024-06-06 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-06

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic pulmonary fibrosis; Remote monitoring; Exacerbation; Prevention
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to assess the feasibility of early detection of acute exacerbations of idiopathic pulmonary fibrosis by the remote monitoring of vital signs.

The main question the study aims to answer is: Could a remote monitoring device allow for earlier detection of exacerbations with individualized monitoring and continuous data collection? All patients will receive conventional clinical follow-up based on their health status and clinical recommendations. At the same time, they will benefit from the Bora Care® medical remote monitoring device.

DETAILED DESCRIPTION:
All patients will receive conventional clinical follow-up based on their health status and clinical recommendations. At the same time, they will benefit from the Bora Care® medical remote monitoring device.

To do this, they will be equipped with a Bora Band® connected wristband that measures vital signs at home, and the Bora Box® Gateway that ensures connectivity and allows automatic data uploading in real time to the Bora Connect® data visualization platform.

The home healthcare provider Air de Bretagne will be involved in the study to support each patient in the use of the connected wristband.

At the end of the follow-up period, the collected data will be retrospectively analysed to identify the most relevant metrics within the time series of vital signs for early detection of Idiopathic Pulmonary Fibrosis exacerbations, and to assess the feasibility of early detection of Idiopathic Pulmonary Fibrosis exacerbations using a score that could trigger an alert prior to the date the patient reports clinical signs or the date the pulmonologist is consulted for exacerbation of Idiopathic Pulmonary Fibrosis.

Procedure:

* Inclusion Visit : 6-minute walk test and prescription of oxygen therapy
* Home Installation Visit: installation of oxygen therapy by Air de Bretagne and setup of the Bora Connect® bracelet and Bora Box® Gateway
* Follow-up Visit with the Pulmonologist at 6 months (M6): routine examinations, satisfaction questionnaire, and quality of life questionnaire
* End of Study Visit with the Pulmonologist at 12 months (M12): routine examinations, satisfaction questionnaire, and quality of life questionnaire.

(In case of exacerbation, the follow-up will be extended by 3 months to collect post-exacerbation data.)

ELIGIBILITY:
Inclusion Criteria:

* Patient over 18 years of age, ideally 50% male and 50% female
* Patient with IPF with a known level of respiratory function (EFR and blood gas less than 3 months)
* Stable patient, i.e. without hospitalisation or exacerbation in the last 3 months
* Patient desaturating at 6MW in ambient air (AA) and requiring ambulatory oxygen therapy (SpO2 AA ⩽ 88%)
* Patient not receiving walking or permanent oxygen therapy at baseline
* Informed patient who has signed consent
* Patient affiliated to a social security scheme
* Patient not monitored by a home healthcare provider other than Air de Bretagne.

Exclusion Criteria:

* Vulnerable patient
* Patient receiving ambulatory or permanent oxygen therapy at baseline
* Patient already seen with another healthcare provider (e.g. OSAS)
* Patient unable to use the Bora Band® tool and without access to a caregiver
* Presence of co-morbidity considered unstable or very severe by the investigator
* Patient protected, under guardianship or incapable of giving free and informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Idiopathic Pulmonary Fibrosis with indication for ambulatory oxygen therapy (Sp02 (peripheral oxygen saturation) ≤ 88% in ambient air during 6-minute walk test)
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Assess the feasibility of early detection of acute IPF exacerbations with the Bora Care® Vital Signs Remote Monitoring Solution. | 1 year
  Correlation between changes in time series of vital signs (heart rate, respiratory rate) in patients in the days prior to diagnosis of exacerbation of Idiopathic Pulmonary Fibrosis and onset of exacerbation of Idiopathic Pulmonary Fibrosis.

SECONDARY OUTCOMES:
Identify relevant metrics in the signals collected by the Bora Care® solution for early detection of medical events. | 1 year
  Evolution of vital signs in patients on days prior to the date of other medical events during follow-up.
Assess compliance with the use of the Bora Care® bracelet by patients. | 1 year
  Number of hours of wearing the Bora Band® bracelet normalised by the total number of hours of the remote monitoring session, information collected via the Bora Care® too.
Assess patient satisfaction and reassurance provided by the remote monitoring solution | 1 year
  Subjective assessment by the patient of the device of the reassurance provided by the device, of the help to resume physical activity provided by the device, obtained using satisfaction questionnaires at M6 and M12.
  SF36 Quality of Life Questionnaire score collected at D0, M6 and M12.
Assess the satisfaction and adherence of healthcare professionals to the remote monitoring solution. | 1 year
  Subjective assessment of health care professionals' satisfaction with and adherence to the Bora Care® remote monitoring solution, including an organizational impact assessment and an assessment of clinical relevance using a questionnaire at the end of the study.
Assess side effects related to the Bora Care® device. | 1 year
  Number and nature of Bora Care® adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Stéphane JOUNEAU, MD, Principal Investigator — CHRU PONTCHAILLOU Rennes
Locations (1):
- Chru Pontchaillou, Rennes, France

IPD SHARING:
Plan to Share IPD: No
Not applicable. Data are not intended to be shared with other researchers.